CLINICAL TRIAL: NCT01235871
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SB1578 When Administered Orally to Healthy Adult Subjects With One Single-Dose Group Crossing Over to Assess Food Effect
Brief Title: A Single and Multiple-Dose Study of SB1578
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SB1578-2010-001
Record Dates: First submitted 2010-11-02; First posted 2010-11-08 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteer
Keywords: Safety; Tolerability; SB1578
MeSH Terms: interventions — 15-(2-(pyrrolidin-1-yl)ethoxy)-7,12,25-trioxa-19,21,24-triazatetracyclo(18.3.1.1(2,5).1(14,18))hexacosa-1(24),2,4,9,14(26),15,17,20,22-nonaene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB1578 (Experimental)
  Interventions: Drug: SB1578
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB1578 — JAK2 Inhibitor
  Arms: SB1578
Drug: Placebo — Control arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of SB1578 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females of non-childbearing potential, 18 to 55 years of age (inclusive).
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55 and 100 kg (inclusive).
* Medically healthy with clinically insignificant screening results.

Exclusion Criteria:

* History or presence of significant disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Assess number of participants with adverse events as a measure of safety and tolerability | 312 hours postdose

SECONDARY OUTCOMES:
Assess pharmacokinetics to determine study drug half-life, maximum concentration time, elimination time, and area under the curve | Predose to 312 hours postdose
Assess pharmacodynamics to determine study drug levels to signal pJAK2, pSTAT3, and pSTAT5 | Predose, 6 and 24 hours postdose
Assess food effects on pharmacokinetics | Predose to 312 hours postdose
Determine recommended dose | March 2011

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Allison, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States